CLINICAL TRIAL: NCT05200065
Title: Prospective Randomized Study Comparing the Intra-operative and Post-operative Outcomes of Bipolar Enucleation of the Prostate Versus Thulium Laser Enucleation
Brief Title: Thulium Laser Versus Bipolar Enucleation of the Prostate
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omar AbdelAziz AbdelHamid, Assistant Lecturer of Urology Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Enucleation techniques for BPH
Record Dates: First submitted 2021-12-14; First posted 2022-01-20 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Benign Prostatic Hyperplasia; Thulium laser enucleation; Bipolar enucleation; Anatomic enucleation of the prostate; Endoscopic Enucleation of the prostate; Thulium laser; Bipolar Plasma energy
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Intervention Model Description: Prospective randomized study comparing two techniques of endoscopic enucleation of the prostate.
Who Masked: Participant
Masking Description: Prospective randomized study comparing the two techniques with patient allocation using computer generated randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thulium Laser Enucleation (Experimental): Patients in this arm will undergo thulium laser enucleation of the prostate.
  Interventions: Procedure: Thulium laser enucleation of the prostate
- Bipolar Enucleation (Experimental): Patients in this arm will undergo bipolar enucleation of the prostate.
  Interventions: Procedure: Bipolar enucleation of the prostate

INTERVENTIONS:
Procedure: Thulium laser enucleation of the prostate — Using the thulium laser to achieve complete endoscopic enucleation of the prostate.
  Arms: Thulium Laser Enucleation
Procedure: Bipolar enucleation of the prostate — Using the bipolar plasma energy to achieve complete endoscopic enucleation of the prostate.
  Arms: Bipolar Enucleation

SUMMARY:
Comparing the peri-operative outcomes in patients with benign prostatic hyperplasia (BPH) who will undergo bipolar enucleation of the prostate versus thulium laser enucleation.

DETAILED DESCRIPTION:
* Benign prostatic hyperplasia (BPH) is one of the most common and bothersome diseases influencing the quality of life of aging males. For decades, transurethral resection of the prostate (TURP) has been recognized as the standard treatment for BPH .Recently, endoscopic laser treatments of BPH has been developed as the result of advances in laser technology and better understanding of tissue-laser interactions and nowadays it represents a challenge for TURP as regards the peri-operative outcomes.
* Both the European Association of Urology (EAU) and American Urological Association (AUA) recommend endoscopic enucleation of the prostate (EEP) as one of the techniques for management of benign prostatic hyperplasia (BPH) with various techniques that could be implemented including enbloc and three/two lobe enucleation.
* The classical laser enucleation technique consists of a three-lobe enucleation of the adenoma with separate enucleation of the median and lateral lobes. Scoffone and Cracco developed an "en-bloc" enucleation technique for HoLEP (holmium laser enucleation) in 2016, showing a potential role to ease some difficult intraoperative steps of enucleation and to improve the learning curve and both of the techniques mentioned were found to be applicable for bipolar endoscopic enucleation as well.
* Regarding the thulium laser physical properties; its wavelength is very close to the peak for absorption in water about 1940 nm being similar to the holmium laser wavelength which is about 2010 nm. However, unlike the pulsed wave holmium laser, this high density energy of thulium laser is best delivered in a continuous wave. This is translated into more efficient vaporization and shallower depth of penetration in tissue, which has been reported to be 0.2 mm as compared with 0.4 mm for holmium lasers. In thulium laser; the continuous wave mode is more suitable for hemostasis and coagulation of tissue, whereas the pulsed mode is more suited for lithotripsy.
* BipolEP (Bipolar enucleation of the prostate) has been performed as an effective method for the management of BPH in some institutions. Bipolar enucleation of prostate is a done using energy source of a bipolar electrosurgical unit. Enucleated prostatic tissues are then removed with a morcellator.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with BPH who are unsatisfied with medical treatment having a Qmax of less than 15 cm/s.
2. Patients with BPH who had refractory retention.
3. Patients with complicated BPH (eg; chronic retention, refractory hematuria, bladder stones).
4. Prostate size of at least 80 grams or more.

Exclusion Criteria:

1. Patients with a bladder mass.
2. Patients with prostate cancer.
3. Patients suffering from a urethral stricture.
4. Patients with previous endoscopic or surgical prostate intervention.
5. Prostate size less than 80 grams.

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Effect on the operative time and other intra-operative and post-operative parameters | 3 to 6 month
  Effect of the chosen technique on the operative time including both enucleation and morcellation times.
  The occurrence of any inta-operative complications including significant blood loss necessitating blood transfusion, capsular perforation, sub-trigonal dissection and complications related to morcellation for example bladder perforation.
  The occurrence of any post-operative complications which is divided into either immediate post-operative and long term complications.
  Immediate post-operative complications occurring in the first 48 hours after enucleation include affection of the hemodynamics and vital signs of the patient, drop in hemoglobin level, high grade fever or uro-sepsis, retention with re-catheterization, hematuria with clot retention.
  long term complications occurring include persistent urge or stress urinary incontinence, secondary hemorrhage with hematuria and clot retention, recurrent urinary tract infections, urethral stricture or bladder neck contracture.

SECONDARY OUTCOMES:
Change of the urine flow of the patients. | 3 to 6 month
  Improvement of the uroflowmetry parameters after catheter removal especially the Qmax (maximum flow rate), Qavg (Average flow rate) in addition to a bell shaped curve in the flowmetry plotted curve.
Change of the IPSS (International Prostatic Symptom Score) of the patients | 3 to 6 month
  Improvement of the IPSS score of the patients after catheter removal compared to the value of the IPSS before enucleation.
  Values of the IPSS:
  Mild Symptoms from 1 to 7 Moderate Symptoms from 8 to 19 Severe Symptoms from 20 to 35
Change of residual urine volume after surgery | 3 to 6 month
  Reduction in the amount of residual urine by US after catheter removal below 150 cc.

CONTACTS AND LOCATIONS:
Overall Officials: Omar AbdelRazzak, MD Urology, Study Director — Kasr AlAiny
Locations (1):
- Kasr AlAiny School of Medicine, Cairo, Egypt

REFERENCES:
- [Background] Berry SJ, Coffey DS, Walsh PC, Ewing LL. The development of human benign prostatic hyperplasia with age. J Urol. 1984 Sep;132(3):474-9. doi: 10.1016/s0022-5347(17)49698-4. PMID 6206240
- [Background] Gravas S, Bachmann A, Reich O, Roehrborn CG, Gilling PJ, De La Rosette J. Critical review of lasers in benign prostatic hyperplasia (BPH). BJU Int. 2011 Apr;107(7):1030-43. doi: 10.1111/j.1464-410X.2010.09954.x. PMID 21438974
- [Background] Enikeev D, Glybochko P, Okhunov Z, Alyaev Y, Rapoport L, Tsarichenko D, Enikeev M, Sorokin N, Dymov A, Taratkin M. Retrospective Analysis of Short-Term Outcomes After Monopolar Versus Laser Endoscopic Enucleation of the Prostate: A Single Center Experience. J Endourol. 2018 May;32(5):417-423. doi: 10.1089/end.2017.0898. Epub 2018 Mar 13. PMID 29430969
- [Background] Scoffone CM, Cracco CM. The en-bloc no-touch holmium laser enucleation of the prostate (HoLEP) technique. World J Urol. 2016 Aug;34(8):1175-81. doi: 10.1007/s00345-015-1741-y. Epub 2015 Dec 11. PMID 26658753
- [Background] Fried NM, Murray KE. High-power thulium fiber laser ablation of urinary tissues at 1.94 microm. J Endourol. 2005 Jan-Feb;19(1):25-31. doi: 10.1089/end.2005.19.25. PMID 15735378
- [Background] Hardy LA, Wilson CR, Irby PB, Fried NM. Thulium fiber laser lithotripsy in an in vitro ureter model. J Biomed Opt. 2014 Dec;19(12):128001. doi: 10.1117/1.JBO.19.12.128001. PMID 25518001
- [Background] Ryang SH, Ly TH, Tran AV, Oh SJ, Cho SY. Bipolar enucleation of the prostate-step by step. Andrologia. 2020 Sep;52(8):e13631. doi: 10.1111/and.13631. Epub 2020 May 22. PMID 32441397